CLINICAL TRIAL: NCT00750282
Title: An Open-label, Non-randomized, Multi-center Study to Optimize Image Assessment and Evaluate the Efficacy and Safety of BAY 94-9172 (ZK 6013443) Positron Emission Tomography (PET) for Detection/Exclusion of Cerebral Amyloid Beta in Patients With Probable Alzheimer's Disease Compared to Healthy Volunteers
Brief Title: Phase II Study of Florbetaben (BAY 94-9172) PET Imaging for Detection/Exclusion of Cerebral β-amyloid in Patients With Probable Alzheimer's Disease Compared to Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 311741; 2007-002256-42 (EudraCT Number); 311741 (Other: company internal)
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer Disease; Amyloid Beta-Protein
Keywords: Alzheimer Disease; Amyloid beta-Protein
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Florbetaben (BAY94-9172) (Experimental)
  Interventions: Drug: Florbetaben (BAY94-9172)

INTERVENTIONS:
Drug: Florbetaben (BAY94-9172) — Healthy volunteers and patients with probable Alzheimer's disease receiving single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions

SUMMARY:
The aim of this study is to evaluate the efficacy, safety of a single dose of BAY 94-9172 (ZK 6013443) as an investigational medicinal product (IMP) in detecting cerebral protein-plaque (amyloid beta) with positron emission tomography (PET). IMP binds to amyloidal beta protein accumulating in brain tissue already from early stages of Alzheimer's disease (AD). IMP is therefore a potential tracer to be used for detecting amyloid plaques. For each subject it is required to visit the study centre during the screening phase, on the PET imaging day and for 1 follow-up visit on the next day. A telephone call for safety follow-up will be performed 7 days after IMP administration. During the screening phase the subject's medical, neurological and surgical history, specific laboratory tests related to AD, MRI of the brain and certain neuro-psychiatric tests will be performed. Clinical safety measures (physical examinations, vital signs, electrocardiogram (ECG) and laboratory tests) will be performed on the PET imaging day before IMP injection and monitored during and after two PET imaging sessions. Clinical safety measures will be performed again on the follow-up visit next day. The results of PET imaging with IMP will be compared between probable AD patients and healthy volunteers (HV). The clinical diagnosis is based on international validated and accepted criteria and established after comprehensive clinical and neuro-psychiatric examinations

ELIGIBILITY:
Inclusion Criteria:

* Each subject / Healthy volunteer (HV) who meets the following criteria will be eligible for enrollment into the study:

  * Is a man or woman and is > 55 of age, whereby females must be without childbearing potential (confirmed by either: age >/= 60; or history of hysterectomy, or last spontaneous bleeding at least 2 years prior to the study start)
  * Has at least 6 years of education
  * Is able to provide informed consent, understand the information provided on the purpose and conduct of the trial and to comply with study procedures
  * Possesses a general health that permits adequate compliance with all study procedures
  * The subject, or the subject and caregiver (for probable AD patients) will be compliant and have a high probability of completing the study
  * Informed consent has been signed and dated (with time) by the subject and/or the subject's caregiver (for probable AD patients)
* Inclusion criteria for HV only:

  * Has no evidence of cognitive impairment
  * Has MRI brain scan that has been judged as "normal" (age- appropriate)
* Inclusion criteria for patients with AD only:

  * Presents with positive assessment for dementia of Alzheimer's type
  * Does not fulfill the criteria Dementia with Lewy Bodies (DLB) or Vascular Dementia (VaD)
  * MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease
  * Has a caregiver that is willing and able to attend all study visits and perform the psychometric tests requiring the presence of a caregiver

Exclusion Criteria:

* Has any contraindication to MRI examination scan
* Is scheduled for surgery and/or another invasive procedure within the time period of up to 24 hours following IMP application
* Is allergic to the IMP or any of its constituents and/or has a history of severe allergic reactions to drugs or allergens (e.g. patients / volunteers with allergic asthma)
* is critically ill and/or medically unstable and whose clinical course during the observation period is unpredictable
* Has a history of exposure to any radiation >15 milli Sieverts (mSv)/year (e.g. occupational or radiation therapy)
* Is receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)
* Has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening, and/or any radiopharmaceutical
* Has a brain tumor or other intracranial lesion, a disturbance of cerebro-spinal fluid (CSF) circulation (e.g., normal pressure hydrocephalus) and/or a history of head trauma or brain surgery
* Has an inflammatory or infectious central nervous system (CNS) disease, e.g. multiple sclerosis, HIV, syphilis, or Creutzfeldt-Jacob disease
* Has a history, physical, laboratory or imaging findings indicative of a neurological or psychiatric illness
* Has another disease that can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function)
* Has a history of alcohol or drug abuse
* Has history of severe persistent depression

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- United States (6):
  - Sun City, Arizona
  - Stanford, California
  - New Haven, Connecticut
  - New York, New York
  - The Bronx, New York
  - Providence, Rhode Island
- Australia (3):
  - Westmead, New South Wales
  - Adelaide, South Australia
  - Heidelberg, Victoria
- Germany (8):
  - Erlangen, Bavaria
  - München, Bavaria
  - Essen, North Rhine-Westphalia
  - Jülich, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Japan (2):
  - Kobe, Hyōgo
  - Bunkyo-ku, Tokyo
- Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Barthel H, Gertz HJ, Dresel S, Peters O, Bartenstein P, Buerger K, Hiemeyer F, Wittemer-Rump SM, Seibyl J, Reininger C, Sabri O; Florbetaben Study Group. Cerebral amyloid-beta PET with florbetaben (18F) in patients with Alzheimer's disease and healthy controls: a multicentre phase 2 diagnostic study. Lancet Neurol. 2011 May;10(5):424-35. doi: 10.1016/S1474-4422(11)70077-1. Epub 2011 Apr 8. PMID 21481640
- [Derived] Bullich S, Roe-Vellve N, Marquie M, Landau SM, Barthel H, Villemagne VL, Sanabria A, Tartari JP, Sotolongo-Grau O, Dore V, Koglin N, Muller A, Perrotin A, Jovalekic A, De Santi S, Tarraga L, Stephens AW, Rowe CC, Sabri O, Seibyl JP, Boada M. Early detection of amyloid load using 18F-florbetaben PET. Alzheimers Res Ther. 2021 Mar 27;13(1):67. doi: 10.1186/s13195-021-00807-6. PMID 33773598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were two parts in this study, Part A and Part B. Part A was conducted in Australia, Germany, Switzerland and USA. Subjects were recruited from 17 centers. HVs were age matched to subjects with probable Alzheimer's (AD).
  Part B was conducted in Australia, Germany, Japan, Switzerland, and USA, subjects recruited from 22 centers.
Pre-assignment Details: Part A screened 214 subjects; 113 AD and 101 HV. There were 63 screen failures (40 for inclusion criteria, 14 withdrew consent, 9 for other reasons) and one dropout prior to receiving study drug.
  Part B screened 392 subjects; 204 AD and 188 HV. There were 118 screen failures for similar reasons and 2 dropouts prior to receiving study drug.
Groups:
- Part A Healthy Volunteers: Florbetaben (BAY94-9172) : Healthy volunteers receiving 300 megabequerel (MBq) single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions.
- Part A Alzheimer Patients; Part B Alzheimer Patients: Florbetaben (BAY94-9172) : Patients with probable Alzheimer's disease receiving 300 MBq single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions
- Part B Healthy Volunteers: Florbetaben (BAY94-9172) : Healthy volunteers receiving 300 MBq single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions
Period: Overall Study
Arm/Group | Part A Healthy Volunteers | Part A Alzheimer Patients | Part B Healthy Volunteers | Part B Alzheimer Patients
Started | 69 | 82 | 126 | 148
Completed | 69 | 81 | 125 | 147
Not Completed | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: 1. dropout in Part A occurred due to pre-treatment AEs.
  2. dropouts in Part B occurred due to withdrawal of consent.
Groups:
- Part A Healthy Volunteers; Part B Healthy Volunteers: Florbetaben (BAY94-9172) : Healthy volunteers receiving single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions
- Total: Total of all reporting groups
Arm/Group | Part A Healthy Volunteers | Part A Alzheimer Patients | Part B Healthy Volunteers | Part B Alzheimer Patients | Total
Number analyzed (Participants) | 69 | 81 | 125 | 147 | 422
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 21 | 15 | 78
  >=65 years | 46 | 62 | 104 | 132 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6.86) | 70.7 (7.82) | 70.7 (6.30) | 73.9 (7.30) | 71.4 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 52 | 73 | 200
  Male | 30 | 45 | 73 | 74 | 222
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 22 | 31 | 64
  Australia | 9 | 6 | 11 | 5 | 31
  Germany | 49 | 71 | 63 | 72 | 255
  Switzerland | 3 | 1 | 0 | 11 | 15
  Japan | 0 | 0 | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Specificity and Sensitivity of Florbetaben PET Scans Obtained in Part A Using Two Separate Algorithms and the Onsite Clinical Diagnosis as the Standard of Truth
Description: Part A: For the calculation of sensitivity/specificity, a patient with probable AD was expected to have a positive florbetaben PET scan which was considered a match for sensitivity. A HV was expected to have a negative florbetaben PET scan which was considered a match for specificity. Standard of truth was the onsite clinical diagnosis.
  Two Beta-Amyloid Plaque Load (BAPL) algorithms for assessing the normality/abnormality of beta-amyloid plaque load in the brain scans were used.
  Using algorithm A (Majority Read), a brain scan of a subject with a BAPL score of "1" (without beta-amyloid plaque load) or "2" (with minor beta-amyloid plaque load) was considered normal and a BAPL score of "3" (with significant beta-amyloid plaque load) was considered abnormal.
  Using algorithm B (Average), a brain scan of a subject with a BAPL score of "1" was considered normal and a brain scan with a BAPL score of "2" or "3" was considered abnormal. Algorithm B was used in Part B and in the final
Time Frame: 90 - 110 min after investigational medical product (IMP) injection
Population: All subjects who had PET imaging data and did not have a major protocol violation were included in the analysis.(n=146)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- AD (Sensitivity) Group: All evaluated subjects with Alzheimer's disease
- HV (Specificity) Group: All evaluated healthy volunteers
Arm/Group | AD (Sensitivity) Group | HV (Specificity) Group
Number analyzed (Participants) | 78 | 68
percentage of subjects
  Majority Read Sens/ Spec (BAPL2 = abnormal) | 79.49 [70.47 to 88.51] | 91.18 [84.38 to 97.97]
  Average Sens / Spec (BAPL2 = normal) | 74.79 [65.69 to 83.88] | 96.08 [91.85 to 100.30]

2. Primary Outcome: Specificity and Sensitivity of Florbetaben PET Scans Obtained in Part B Using Two Separate Algorithms and the Onsite Clinical Diagnosis as the Standard of Truth.
Description: Part B: For the calculation of sensitivity/specificity, a patient with probable AD was expected to have a positive florbetaben PET scan, ie,abnormal scan (BAPL scores "2" or "3") which was considered a match for sensitivity. A HV was expected to have a negative florbetaben PET scan, ie,normal scan (BAPL score "1") which was considered a match for specificity.
  The clinical diagnosis was established by an independent consensus panel (CP) of experts in dementia.
  Two independent sets of PET data reads were performed. The first set was performed by a panel of three readers who received live, instructor-led training on the visual assessment procedure. The second set was performed by a panel of five separate readers who were trained on the visual assessment procedure with electronic media.
Time Frame: 90 - 110 min after IMP injection
Population: All subjects who had PET imaging data and did not have a major protocol violation were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- AD (Sensitivity) Group: All subjects evaluated as probable AD by consensus panel
- HV (Specificity) Group: All subjects evaluated as healthy volunteer by consensus panel
Arm/Group | AD (Sensitivity) Group | HV (Specificity) Group
Number analyzed (Participants) | 116 | 118
percentage of subjects
  Sens / Spec (average 3 readers) | 67.24 [58.70 to 75.78] | 96.61 [93.34 to 99.88]
  Sens / Spec (additional read, median 5 readers) | 78.5 [71.0 to 85.9] | 89.2 [83.6 to 94.7]

3. Secondary Outcome: Sensitivity and Specificity for All Participants Using Two Additional Imaging Windows for the Visual Assessment
Description: PET scans from two additional imaging windows (45-60 min and 110-130 min) were visually assessed
Time Frame: 45 - 60 min and 110 - 130 min after IMP injection
Population: All subjects who had PET imaging data and did not have a major protocol violation were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- AD (Sensitivity) Group (Part A): All evaluated subjects with Alzheimer's disease from Part A
- HV (Specificity) Group (Part A): All evaluated healthy volunteers from Part A
- AD (Sensitivity) Group (Part B): All evaluated subjects with probable Alzheimer's disease from part B
- HV (Specificity) Group (Part B): All evaluated healthy volunteers from Part B
Arm/Group | AD (Sensitivity) Group (Part A) | HV (Specificity) Group (Part A) | AD (Sensitivity) Group (Part B) | HV (Specificity) Group (Part B)
Number analyzed (Participants) | 78 | 68 | 116 | 118
percentage of subjects
  Sensitivity & Specificity (45-60 min) | 73.93 [64.88 to 82.98] | 94.61 [90.36 to 98.85] | 71.55 [63.34 to 79.76] | 94.07 [89.81 to 96.55]
  Sensitivity & Specificity (110-130 min) | 70.56 [60.98 to 80.15] | 98.01 [95.65 to 100.37] | 73.04 [64.93 to 81.15] | 96.58 [93.29 to 99.87]

4. Secondary Outcome: Kappa Coefficient as a Measure of Agreement Between Readers Concerning the Visual Assessment of Abnormality of the Brain Scan (Based on BAPL Score)
Description: The agreement between 3 blinded readers concerning the visual assessment of abnormality of the brain scan (based on BAPL score) was measured by the kappa coefficient. Kappa values close to 1.0 indicate a high agreement while values close to 0 indicate random agreement.
Time Frame: 45-60 min, 90-110 min, 110-130 min
Population: All subjects who had PET imaging data and did not have a major protocol violation were included in the analysis
Measure: Number; unit: Kappa coefficient
Groups:
- Imaging Window 45-60 Min Part A: Kappa coefficient estimate for PET data collected 45-60 min post-injection in Part A
- Imaging Window 90-110 Min Part A: Kappa coefficient estimate for PET data collected 90-110 min post-injection in Part A
- Imaging Window 110-130 Min Part A: Kappa coefficient estimate for PET data collected 110-130 min post-injection in Part A.
- Imaging Window 45-60 Min Part B: Kappa coefficient estimate for PET data collected 45-60 min post-injection in Part B
- Imaging Window 90-110 Min Part B: Kappa coefficient estimate for PET data collected 90-110 min post-injection in Part B
- Imaging Window 110-130 Min Part B: Kappa coefficient estimate for PET data collected 110-130 min post-injection in Part B.
Arm/Group | Imaging Window 45-60 Min Part A | Imaging Window 90-110 Min Part A | Imaging Window 110-130 Min Part A | Imaging Window 45-60 Min Part B | Imaging Window 90-110 Min Part B | Imaging Window 110-130 Min Part B
Number analyzed (Participants) | 150 | 150 | 150 | 272 | 272 | 272
Kappa coefficient | 0.56 | 0.60 | 0.67 | 0.78 | 0.86 | 0.86

5. Secondary Outcome: Standard Uptake Value Ratios for Florbetaben Signal
Description: The Standard Uptake Value Ratios for florbetaben signal in the frontal cortex, lateral temporal cortex, parietal cortex, anterior cingulate, posterior cingulate cortex, occipital cortex, and cerebellum (white matter) were determined as a quantitative measure of tracer uptake. The SUV is defined as the ratio of (1) the tissue radioactivity concentration c (in MBq/kg) at time point t, and (2) the injected activity (in MBq, extrapolated to the same time t) divided by the body weight (in kg). These SUV numbers from regions of interest were then used to derive SUV ratios (SUVR) using the SUV from the cerebellar cortex as reference.)
Time Frame: 90-110 min post injection
Population: All subjects who had PET imaging data and did not have a major protocol violation were included in the analysis
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Alzheimer's (AD) Group (Part A): All evaluated subjects with Alzheimer's disease
- Healthy Volunteer (HV) Group (Part A): All evaluated healthy volunteers
- Alzheimer's (AD) Group (Part B): All subjects with consensus panel based diagnosis of "probable AD"
- Healthy Volunteer (HV) Group (Part B): All subjects that were confirmed by consensus panel as healthy volunteers
Arm/Group | Alzheimer's (AD) Group (Part A) | Healthy Volunteer (HV) Group (Part A) | Alzheimer's (AD) Group (Part B) | Healthy Volunteer (HV) Group (Part B)
Number analyzed (Participants) | 78 | 68 | 116 | 118
ratio
  Frontal cortex | 1.608 (0.3207) [61.47 to 78.18] | 1.295 (0.1151) [86.50 to 96.55] | 1.646 (0.2905) | 1.301 (0.1961)
  Lateral temporal cortex | 1.571 (0.2881) [51.44 to 69.25] | 1.259 (0.1058) [92.13 to 99.40] | 1.619 (0.2787) | 1.292 (0.1620)
  Parietal cortex | 1.528 (0.2896) [65.22 to 81.33] | 1.234 (0.1161) [87.58 to 97.16] | 1.602 (0.2705) | 1.267 (0.1709)
  Anterior cingulate | 1.723 (0.3522) [63.34 to 79.76] | 1.397 (0.1425) [89.81 to 98.33] | 1.786 (0.3145) | 1.434 (0.2387)
  Posterior cingulate cortex | 1.795 (0.3149) [66.85 to 82.72] | 1.422 (0.1565) [90.87 to 98.87] | 1.852 (0.3187) | 1.493 (0.2351)
  Occipital cortex | 1.495 (0.2203) | 1.309 (0.0864) | 1.560 (0.2460) | 1.341 (0.1281)
  Composite SUVR | 1.620 (0.29) | 1.320 (0.11) | 1.678 (0.2699) | 1.355 (0.1784)

ADVERSE EVENTS:
Time Frame: A maximum of 64 days. Up to 56 days during the screening process and 8 days from baseline to second follow-up visit.
Groups:
- Part A Healthy Volunteers; Part B Healthy Volunteers: Florbetaben (BAY94-9172) : Patients with probable Alzheimer's disease receiving single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions
- Part A Alzheimer Patients; Part B Alzheimer Patients: Florbetaben (BAY94-9172) : Healthy volunteers receiving single injection of investigational medicinal product BAY 94-9172 followed by subsequent PET imaging sessions
Arm/Group | Part A Healthy Volunteers | Part A Alzheimer Patients | Part B Healthy Volunteers | Part B Alzheimer Patients
Serious Adverse Events (participants affected / at risk) | 1/69 | 1/81 | 2/125 | 0/147
Other Adverse Events (participants affected / at risk) | 10/69 | 3/81 | 17/125 | 23/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Healthy Volunteers (N=69) | Part A Alzheimer Patients (N=81) | Part B Healthy Volunteers (N=125) | Part B Alzheimer Patients (N=147)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Clear cell endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Healthy Volunteers (N=69) | Part A Alzheimer Patients (N=81) | Part B Healthy Volunteers (N=125) | Part B Alzheimer Patients (N=147)
Application site erythema (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (6)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 2 (2) | 8 (8)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 7 (8) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less